CLINICAL TRIAL: NCT07405216
Title: Efficacy and Safety of Sodium-Glucose Cotransporter-2 Inhibitors in Adolescents With Persistent Albuminuria: A Randomized Controlled Clinical Trial
Brief Title: Efficacy and Safety of Sodium-Glucose Cotransporter-2 Inhibitors in Adolescents With Early Stages of Chronic Kidney Disease
Acronym: IECA-MEX
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centenario Hospital Miguel Hidalgo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INAER2026-1
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Chronic Kidney Disease (Mild to Moderate); Albuminuria; Adolescent; Sodium Glucose Co-Transporter 2 Inhibitors
Keywords: Chronic kidney disease; Persistent albuminuria; sodium glucose co-transporter 2 inhibitors
MeSH Terms: conditions — Renal Insufficiency, Chronic; Albuminuria | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Adolescents with persistent albuminuria
  Interventions: Drug: Dapagliflozin (10mg Tab)
- Control group (Placebo Comparator): Placebo 10 mg daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin (10mg Tab) — Dapagliflozin 10 mg daily
  Arms: Intervention
Drug: Placebo — Placebo 10 mg daily
  Arms: Control group

SUMMARY:
Chronic kidney disease (CKD) is highly prevalent in the state of Aguascalientes, Mexico, particularly among adolescents and young adults. Epidemiologic and histologic studies suggest that this burden is largely driven by reduced nephron endowment of prenatal origin, leading to compensatory glomerular hyperfiltration, adaptive podocytopathy, and persistent albuminuria at early stages of disease.

Sodium-glucose cotransporter-2 inhibitors (SGLT2i) have demonstrated nephroprotective effects in adult populations with CKD, including reductions in albuminuria and slowing of disease progression, independent of diabetes status. However, no randomized controlled trials have evaluated the efficacy and safety of SGLT2 inhibitors in adolescents with early-stage CKD and persistent albuminuria.

This randomized, double-blind, placebo-controlled clinical trial aims to evaluate whether treatment with an SGLT2 inhibitor reduces albuminuria in adolescents aged 14 to 18 years with persistent microalbuminuria (albumin-to-creatinine ratio 30-300 mg/g) and preserved kidney function. Participants will be randomized in a 2:1 ratio to receive dapagliflozin 10 mg daily or placebo for six months. The primary outcome is the change in urinary albumin-to-creatinine ratio from baseline to six months. Secondary outcomes include changes in estimated glomerular filtration rate and safety outcomes.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a major global health problem and represents one of the fastest-growing causes of mortality worldwide. In the state of Aguascalientes, Mexico, CKD prevalence is among the highest reported globally, with an unusually high burden affecting adolescents and young adults.

Statewide screening programs and renal biopsy registries have identified a distinct epidemiologic and histologic pattern in this region. Adolescents with early-stage CKD frequently present with persistent albuminuria, glomerulomegaly, absence of interstitial fibrosis, and adaptive podocytopathy, findings consistent with reduced nephron endowment of prenatal origin. Over time, these lesions may progress to adaptive focal segmental glomerulosclerosis and clinically significant CKD in young adulthood. The predominant pathogenic mechanism in this population is believed to be glomerular hyperfiltration.

Pharmacologic therapies targeting hyperfiltration have proven efficacy in slowing CKD progression. Renin-angiotensin-aldosterone system inhibitors are standard of care, and more recently, sodium-glucose cotransporter-2 inhibitors have demonstrated substantial nephroprotective effects in adult populations, including patients without diabetes and across a wide range of albuminuria levels. Despite this evidence, adolescents and patients with early-stage CKD (G1-G2 A2) have been systematically excluded from major randomized trials.

This study is a randomized, double-blind, placebo-controlled clinical trial designed to evaluate the efficacy and safety of an SGLT2 inhibitor in adolescents with persistent albuminuria and preserved kidney function. Eligible participants are adolescents aged 14 to 18 years residing in Aguascalientes with persistent microalbuminuria (albumin-to-creatinine ratio 30-300 mg/g), estimated glomerular filtration rate ≥60 mL/min/1.73 m², and no identifiable secondary cause of kidney disease.

After screening and baseline evaluation-including medical history, laboratory testing, immunologic studies, and renal ultrasound-eligible participants will be randomized in a 2:1 ratio to receive dapagliflozin 10 mg daily or matching placebo for a total duration of six months. All participants will receive standardized nutritional counseling.

Follow-up visits will occur every two months and will include clinical assessment, physical examination, blood pressure measurement, and laboratory testing. Urinary albumin-to-creatinine ratio will be measured using standardized laboratory methods.

The primary endpoint is the change in urinary albumin-to-creatinine ratio from baseline to six months, analyzed using log-transformed values. Secondary endpoints include changes in estimated glomerular filtration rate and assessment of safety outcomes, including adverse events such as hypotension and urinary tract infections.

This trial seeks to generate high-quality evidence on the efficacy and safety of SGLT2 inhibitors in adolescents with early-stage CKD, a population with a disproportionate disease burden and limited therapeutic evidence.

ELIGIBILITY:
Inclusion Criteria:Age 14-18 years

Residence in Aguascalientes

Persistent albuminuria (ACR >30 and <300 mg/g)

Estimated glomerular filtration rate ≥60 mL/min/1.73 m²

No identifiable secondary cause (e.g., lupus, diabetes mellitus)

Renal biopsy showing adaptive podocytopathy or perihilar focal segmental glomerulosclerosis -

Exclusion Criteria:

Hypoalbuminemia

Nephrotic syndrome

Persistent macroalbuminuria (ACR >300 mg/g)

Secondary causes of CKD, including congenital anomalies of the kidney and urinary tract or polycystic kidney disease -

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Albuminuria | 2, 4 and 6 months
  The urinary albumin-to-creatinine ratio (ACR) will be calculated. The primary endpoint will be the log-transformed difference between baseline and six-month ACR. Absolute and relative (% reduction) changes in ACR will also be reported.

SECONDARY OUTCOMES:
Glomerular filtration rate | 2,4 and 6 months
  Glomerular filtration rate estimated with Chronic Kidney Disease in Children under (age) 25 (CKiD U25) equation

OTHER OUTCOMES:
Safety outcomes | 2,4 and 6 months
  Adverse events such as hypotension and urinary tract infections.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 20. Agarwal R, Green JB, Heerspink HJL, et al. Finerenone with Empagliflozin in Chronic Kidney Disease and Type 2 Diabetes. N Engl J Med. 2025;393(6):533-543. doi:10.1056/NEJMoa2410659
- [Background] 19. Kanbay M, Copur S, Bakir CN, Covic A, Ortiz A, Tuttle KR. Glomerular hyperfiltration as a therapeutic target for CKD. Nephrol Dial Transplant. 2024;39(8):1228-1238. doi:10.1093/ndt/gfae027
- [Background] 18. Staplin N, Roddick AJ, Neuen BL, et al. Effects of Sodium Glucose Cotransporter 2 Inhibitors by Diabetes Status and Level of Albuminuria: A Meta-Analysis. JAMA. Published online November 7, 2025. doi:10.1001/jama.2025.20835
- [Background] 17. Heerspink HJL, Stefánsson BV, Correa-Rotter R, et al. Dapagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2020;383(15):1436-1446. doi:10.1056/NEJMoa2024816
- [Background] 16. The EMPA-KIDNEY Collaborative Group, Herrington WG, Staplin N, et al. Empagliflozin in Patients with Chronic Kidney Disease. N Engl J Med. 2023;388(2):117-127. doi:10.1056/NEJMoa2204233
- [Background] 15. KDIGO CKD Work Group. KDIGO 2024 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease. Kidney International. 2024 Apr;105(4S):S117-S314. doi: 10.1016/j.kint.2023.10.018
- [Background] 14. Ortiz A, Arreola Guerra JM, Chan JCN, et al. Preventing chronic kidney disease and maintaining kidney health: conclusions from a Kidney Disease: Improving Global Outcomes (KDIGO) Controversies Conference. Kidney Int. 2025;108(4):555-571. doi:10.1016/j.kint.2025.04.005
- [Background] 13. Alcalde-Ortiz ML, Jaramillo-Arriaga F, Ibarra-Orenday D, et al. Pediatric kidney dimensions and risk of persistent albuminuria in Mexican adolescents. Kidney Int. 2024;105(4):824-834. doi:10.1016/j.kint.2023.11.034
- [Background] 12. Macias Diaz DM, Corrales Aguirre MDC, Reza Escalera AL, et al. Histologic characterization and risk factors for persistent albuminuria in adolescents in a region of highly prevalent end-stage renal failure of unknown origin. Clin Kidney J. 2022;15(7):1300-1311. Published 2022 Jan 14. doi:10.1093/ckj/sfac018
- [Background] 11. United States Renal Data System. 2024 USRDS Annual Data Report: Epidemiology of kidney disease in the United States. National Institutes of Health, National Institute of Diabetes and Digestive and Kidney Diseases, Bethesda, MD, 2024.
- [Background] 10. Registro Estatal Únicio de Enfermedad Renal Crónica del Estado de Aguascalientes. Instituto de Servicios de Salud del Estado de Aguascalientes. https://www.issea.gob.mx/ercpub/en/RepPrevalenciaErcPbiPubV2.asp Date: January 11, 2026
- [Background] 9. Garcia-Garcia G, Gutiérrez-Padilla A, Perez-Gomez HR, et al. Chronic kidney disease of unknown cause in Mexico: The case of Poncitlan, Jalisco. Clin Nephrol. 2020;93(1):42-48. doi:10.5414/CNP92S107
- [Background] 8. Gutierrez-Peña M, Zuñiga-Macias L, Marin-Garcia R, et al. High prevalence of end-stage renal disease of unknown origin in Aguascalientes Mexico: role of the registry of chronic kidney disease and renal biopsy in its approach and future directions. Clin Kidney J. 2021;14(4):1197-1206. doi:10.1093/ckj/sfaa229
- [Background] 7. Barquera S, Hernández-Barrera L, Trejo-Valdivia B, Shamah T, Campos-Nonato I, Rivera-Dommarco J. Obesidad en México, prevalencia y tendencias en adultos. Ensanut 2018-19 [Obesity in Mexico, prevalence andtrends in adults. Ensanut 2018-19.]. Salud Publica Mex. 2020;62(6):682-692. doi:10.21149/11630
- [Background] 6. Arreola-Guerra JM, Martinez-Martinez JI, Multifactorial chronic kidney disease, Nephrology Dialysis Transplantation, 2025;, gfaf122, https://doi.org/10.1093/ndt/gfaf122
- [Background] 5. GBD 2023 Chronic Kidney Disease Collaborators. Global, regional, and national burden of chronic kidney disease in adults, 1990-2023, and its attributable risk factors: a systematic analysis for the Global Burden of Disease Study 2023. Lancet. 2025;406(10518):2461-2482. doi:10.1016/S0140-6736(25)01853-7
- [Background] 4. Francis A, Harhay MN, Ong ACM, et al. Chronic kidney disease and the global public health agenda: an international consensus. Nat Rev Nephrol. 2024;20(7):473-485. doi:10.1038/s41581-024-00820-6
- [Background] 3. Institute for Health Metrics and Evaluation. Global Burden of Disease 2019. Accessed February 14, 2023. https://vizhub.healthdata.org/gbdcompare/
- [Background] 2. GBD 2015 Mortality and Causes of Death Collaborators. Global, regional, and national life expectancy, all-cause mortality, and cause-specific mortality for 249 causes of death, 1980-2015: a systematic analysis for the Global Burden of Disease Study 2015 Lancet. 2016;388(10053):1459-1544. doi:10.1016/S0140-6736(16)31012-1
- [Background] 1. GBD 2023 Chronic Kidney Disease Collaborators. Global, regional, and national burden of chronic kidney disease in adults, 1990-2023, and its attributable risk factors: a systematic analysis for the Global Burden of Disease Study 2023. Lancet. 2025;406(10518):2461-2482. doi:10.1016/S0140-6736(25)01853-7